CLINICAL TRIAL: NCT01088724
Title: Fludarabine, Cyclophosphamide, Doxorubicin and Rituximab for the Treatment of Post-transplant Lymphoproliferative Disease (PTLD)
Acronym: FCD-R
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Responsible Party: Eugenia Giraldi, Ospedali Riuniti di Bergamo, Italy
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: OORRPED 1
Record Dates: First submitted 2010-03-11; First posted 2010-03-17 (Estimated); Last update posted 2010-03-17 (Estimated); Status verified 2010-03

CONDITIONS: Post-transplant Lymphoproliferative Disease (PTLD); Non Burkitt
MeSH Terms: interventions — fludarabine; Cyclophosphamide; Doxorubicin; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- chemotherapy (Experimental)
  Interventions: Drug: fludarabine, cyclophosphamide, doxorubicin, rituximab

INTERVENTIONS:
Drug: fludarabine, cyclophosphamide, doxorubicin, rituximab — Fludarabine i.v.(30 mg/sqm/day,day 1,2,3); Cyclophosphamide i.v.(750 mg/sqm, day 1); Doxorubicin i.v.(30 mg/sqm, day 1); Rituximab i.v. (375 mg/sqm, day 4).

SUMMARY:
Fludarabine may be of benefit to prevent rejection of grafted solid organs in children during chemo-immunotherapy treatment for post transplant lymphoproliferative diseases (PTLDs).

DETAILED DESCRIPTION:
Eligible to this study were patients less than 18 years old, presenting with non Burkitt, aggressive, CD20 positive PTLD, after solid organ transplants.

Induction therapy consisted of two cycles of a combination of Fludarabine(30mg/sqm/day, days 1,2,3), Cyclophosphamide (750 mg/sqm/day, day 1), Doxorubicin (30 mg/sqm/day, day 1)and Rituximab (375 mg/sqm/day, day 4).

Thereafter consolidation therapy was given as follows: two blocks for stage II or III with LDH less than 500 IU/L; three blocks for stage III with LDH >500 and < 1000 IU/L or stage IV with LDH < 1000 IU/L; four blocks for stage III or IV with LDH > 1000 IU/L. Blocks given were modified BFM blocks used for treatment of non Hodgkin B-lymphomas, as follows:

Block 1: High Dose Methotrexate (HDMTX) 1.5 gr/sqm; Vincristine (VCR,1.5 mg/sqm); Cytarabine (from 120 to 150 mg/sqm x4); Ifosfamide (600 mg/sqm/day x5); VP-16 (80 mg/sqm/day x2); Dexamethasone (DXM,10 mg/sqm/day for 5 ays); Intrathecal Methotrexate-Cytarabine-Methylprednisolone(TIT).

Block 2:HDMTX (3 gr/sqm); VCR (1.5 mg/sqm); Daunomycin (20 mg/sqm/day x2); Cyclophosphamide (160 mg/sqm/day x5); DXM (10 mg/sqm/day x5); TIT

Block 3:Vindesine (3 mg/sqm); Cytarabine (3000 mg/sqm q 12 hours x4); VP-16 (100 mg/sqm q 12 hours x4); DXM (20 mg/sqm/day x5);

Block 4 as Block 1.

Outcome measures are: achievement of complete remission after induction therapy; incidence of infectious episodes; neurological toxicity; incidence of graft rejection; duration of complete remission.

ELIGIBILITY:
Inclusion Criteria:

* Children less 18 years old and
* Non Burkitt, CD20 positive aggressive PTLD and
* Solid organ transplant

Exclusion Criteria:

* Burkitt PTLD

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2002-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Complete remission rate | 6 months
  No evidence of disease
graft rejection rate | 1 year after treatment
  preservation of normal organ function

SECONDARY OUTCOMES:
Continuous complete remission rate | five years after the diagnosis
  No evidence of disease

CONTACTS AND LOCATIONS:
Overall Officials: Valentino Conter, MD, Study Chair — Department of Pediatrics, Ospedali Riuniti di Bergamo
Locations (1):
- Ospedali Riuniti di Bergamo, Bergamo, BG, Italy